CLINICAL TRIAL: NCT04715776
Title: Supplementation of Brown Seaweed on Insulin Resistance of NAFLD Patients With Pre- or Type 2-Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Hi-Q Marine Biotech International, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N201805009
Record Dates: First submitted 2018-09-04; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-08

CONDITIONS: Type II Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-DM patients with placebo (Placebo Comparator): Pre-Diabetes patients uptake placebo as dietary supplement
  Interventions: Dietary Supplement: placebo
- Pre-DM patients with supplement (Experimental): Pre-Diabetes patients uptake Brown seaweed as dietary supplement
  Interventions: Dietary Supplement: Brown seaweed
- DM patients with placebo (Placebo Comparator): Diabetes patients uptake placebo as dietary supplement.
  Interventions: Dietary Supplement: placebo
- DM patients with supplement (Experimental): Diabetes patients uptake Brown seaweed as dietary supplement
  Interventions: Dietary Supplement: Brown seaweed

INTERVENTIONS:
Dietary Supplement: Brown seaweed — Uptake of 1650 mg brown seaweed product twice daily
  Arms: DM patients with supplement; Pre-DM patients with supplement
Dietary Supplement: placebo — Uptake of 1650 mg placebo twice daily
  Arms: DM patients with placebo; Pre-DM patients with placebo

SUMMARY:
Investigators research team conducted a previous human clinical trial of brown algae and conducted liver and metabolic indicators of brown algae to improve nonalcoholic fatty liver disease, and found brown algae extract (LMF-HSFx, commodity In addition to reducing the liver function index, HbA1c in some patients with early stage diabetes or type 2 diabetes has an improved effect. In the mouse model of type 2 diabetes, comprehensive anti-hyperglycemia, anti-hyperlipidemia and hepatoprotective activity were studied using LMF-HSFx. Intake of LMF-HSFx reduced fasting blood glucose, increased adiponectin levels, reduced urine glucose, and improved hepatic glucose metabolism. LMF-HSFx can improve glucose and lipid metabolism in adipose tissue of diabetic mice, and inflammatory factors such as TNF-α and IL-6 can also be reduced.

In this study,participants will be given Fuco-HiQ, and their effects on blood glucose and various metabolic indicators will be evaluated.

DETAILED DESCRIPTION:
Brown seaweeds rich in flavonoids and bioactive polysaccharides have been shown the potential effects on suppressing fat accumulation, oxidative stress and inflammation in liver. The refined seaweed compounds such as low-molecular-weight-fucoidan (LMF) and high stability fucoxanthin (HSFx), have not been well studied for its biological function.

The high stability fucoxanthin (HSFx) and the low-molecular-weight fucoidan (LMF) were produced by HiQ Marine Biotech Company in Taiwan. Study use fucoidan-fucoxanthin mixture (abbreviated as LMF-HSFx, each capsule contains 275 mg LMF and 275 mg HSFx).

Insulin resistance has a high correlation with fatty liver. Our research team conducted a previous human clinical trial of brown algae and conducted liver and metabolic indicators of brown algae to improve nonalcoholic fatty liver disease, and found brown algae extract (LMF-HSFx, commodity In addition to reducing the liver function index, HbA1c in some patients with early stage diabetes or type 2 diabetes has an improved effect. In the mouse model of type 2 diabetes, comprehensive anti-hyperglycemia, anti-hyperlipidemia and hepatoprotective activity were studied using LMF-HSFx. Intake of LMF-HSFx reduced fasting blood glucose, increased adiponectin levels, reduced urine glucose, and improved hepatic glucose metabolism. LMF-HSFx can improve glucose and lipid metabolism in adipose tissue of diabetic mice, and inflammatory factors such as TNF-α and IL-6 can also be reduced.

Based on these studies, we hope to further explore whether LMF-HSFx can improve insulin resistance and thus assist blood glucose control.In this study,subjects will be given Fuco-HiQ, and their effects on blood glucose and various metabolic indicators will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 20 and 75 years old, biochemical test data and abdominal ultrasound screening were selected according to the following conditions.

1. Prediabetes: AC at 101 to 125 and HbA1c at 5.8 to 6.4 and abdominal ultrasound confirmed fatty liver.
2. Type 2 Diabetes: Abdominal ultrasound confirms the presence of fatty liver; Hypoglycemic agent HbA1c controls 8% (but does not contain Pioglitazone or injection of Liraglutide), or patient HbA1c is controlled below 9% but does not want to increase drug Dosage or add other hypoglycemic agents.

Exclusion Criteria:

1. Severe renal insufficiency (diabetic or eGFR less than 30 mL/min/1.73 m2), severe heart failure (NYHA function classification III or IV), etc.
2. Allergies to seafood and seaweed ingredients.
3. Cannot or refuse to sign test consent.
4. Inject insulin or Liraglutide or take Pioglitazone.
5. Type 1 diabetes patients.
6. People who drink alcohol and take weight-related drugs and health products.
7. There are blood transfusion recipients within three months.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
From baseline to 3 months after using dietary supplements (compare yourself with yourself), follow up for a total of 12 months | 12 months
  The change of HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shun Wu, Study Director — Taipei Municipal Wanfang Hospital
Locations (1):
- Wanfang Hospital, Taipei, Wenshan District, Taiwan